CLINICAL TRIAL: NCT00328783
Title: A Pilot Study Investigating Active Breathing Coordinator (ABC) to Reduce Radiation Dose to Normal Structures in Breast Cancer Patients
Brief Title: Using the Active Breathing Control Device to Reduce Radiation Side Effects to Critical Structures in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 02U.282; 2002-31 (Other: CCRRC); JT 1005 (Other: JeffTrial Number)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Active Breathing Control; Active Breathing Coordinator; ABC
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Breathing Coordinator (Experimental): Patients breathe through the ABC device
  Interventions: Device: Active Breathing Coordinator (ABC); Radiation: Radiation Therapy

INTERVENTIONS:
Device: Active Breathing Coordinator (ABC) — The generated dose distributions from the free-breathing versus ABC plans will be compared to assess the volume of normal tissue, as well as target volume irradiated, utilizing dose-volume histograms.
  Other Names: ABC
Radiation: Radiation Therapy

SUMMARY:
The purpose of this study is to evaluate the use of a device that helps coordinate the breathing cycle in the radiation treatment of the breast in order to minimize the radiation dose to the normal structures around the breast.

DETAILED DESCRIPTION:
The Active Breathing Coordinator (ABC) allows for temporary and reproducible immobilization of internal thoracic structures by monitoring the patient's breathing cycle and implementing a breath hold at a predefined lung volume level. While ABC is FDA approved and commercially available, only preliminary dosimetric data is available on a small number of patients with breast cancer. There is some data using ABC for intrathoracic malignancies, which shows that it is feasible and safe to use. ABC can be used to optimize the distance between chest wall, heart and liver. This allows adequate treatment of the breast and underlying chest wall while minimizing irradiated cardiac and liver volume.

ELIGIBILITY:
Inclusion Criteria:

* Requiring adjuvant or post mastectomy radiation therapy with tangential fields or 3-fields
* Adequate pulmonary function
* Presence of 5 cc of the heart or liver with the simulation fields
* Karnofsky Performance Status (KPS) equal to or greater than 70

Exclusion Criteria:

* Pregnant women
* Patients who have had previous ipsilateral breast or thoracic radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pramila Rani Anne, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Breathing Coordinator: Patients breathe through the ABC device
  Active Breathing Coordinator (ABC) : The generated dose distributions from the free-breathing versus ABC plans will be compared to assess the volume of normal tissue, as well as target volume irradiated, utilizing dose-volume histograms.
Period: Overall Study
Arm/Group | Active Breathing Coordinator
Started | 112
Completed | 86
Not Completed | 26
Not completed — Could not tolerate ABC | 21
Not completed — No heart in RT field | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active Breathing Coordinator
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.19 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Dosimetric Evaluation Magnitude of Reduction in Irradiated Normal Tissues
Description: To evaluate the magnitude of reduction in irradiated normal tissues (heart and lung) when using the Active Breathing Coordinator (ABC) in breast patients, as compared to standard, free-breathing.
  The generated dose distributions from the free-breathing vs. ABC plans will be compared to assess the volume of normal tissue, as well as target volume irradiated, utilizing dose-volume histograms. Specifically, for the heart, the volume receiving 55 and 40 Gy will be evaluated; for the liver the volume receiving 50 and 36 Gy, and for the lung, the volume receiving 20 Gy. For the contralateral breast the volume receiving 20 Gy, 30 Gy and 50 Gy will be evaluated. Patients will be treated with the ABC device if there is at least 5 % relative reduction in the volume of a normal tissue irradiated to prescription dose.
Time Frame: At time of radiation
Measure: Mean (95% Confidence Interval); unit: Gy
Arm/Group | Active Breathing Coordinator
Number analyzed (Participants) | 86
Gy
  Free breathing (heart) | 3.0 [2.6 to 3.3]
  ABC (heart) | 1.1 [0.9 to 1.3]
  Free breathing (lung) | 6.0 [5.3 to 6.8]
  ABC (lung) | 5.4 [4.9 to 5.9]

2. Primary Outcome: Proportion of Patients With Reduction in Radiation
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Active Breathing Coordinator
Number analyzed (Participants) | 86
proportion of patients
  5% reduction (heart) | 0.94 [0.86 to 0.98]
  20% reduction (heart) | 0.88 [0.78 to 0.95]
  5% reduction (lung) | 0.56 [0.41 to 0.70]
  20% reduction (lung) | 0.35 [0.22 to 0.49]

3. Secondary Outcome: Toxicity Evaluation
Description: Number of participants that experienced grade three toxicity or higher as a result of treatment.
Time Frame: 30 days post-treatment
Measure: Count of Participants; unit: Participants
Groups:
- Active Breathing Coordinator: Patients breathe through the ABC device
  Active Breathing Coordinator (ABC): The generated dose distributions from the free-breathing versus ABC plans will be compared to assess the volume of normal tissue, as well as target volume irradiated, utilizing dose-volume histograms.
  Radiation Therapy
Arm/Group | Active Breathing Coordinator
Number analyzed (Participants) | 86
Participants | 0

4. Secondary Outcome: Change in Organs at Risk (OAR) Dosimetric Paramaters
Description: To evaluate the magnitude of change in Mean Heart Dose (MHD) and Left lung dose when using the Active Breathing Coordinator (ABC) in breast patients, as compared to standard, free-breathing.
Time Frame: 30 days post-treatment
Measure: Mean (95% Confidence Interval); unit: Gy
Arm/Group | Active Breathing Coordinator
Number analyzed (Participants) | 86
Gy
  Free Breathing (heart) | 2.7 [2.3 to 3.1]
  ABC (Heart) | .88 [0.78 to 0.95]
  Free Breathing (Lung) | 6.4 [5.7 to 7.0]
  ABC (Lung) | .31 [.20 to .43]

5. Secondary Outcome: Number of Participants With Toxicity of Treatment of Adjuvant Radiotherapy for Breast Cancer With the ABC Device.
Description: To monitor the toxicity of treatment of adjuvant radiotherapy for breast cancer with the ABC device.
Time Frame: 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Breathing Coordinator
Number analyzed (Participants) | 86
Participants
  Acute skin and soft tissue toxicity : Grade 1 | 59
  Acute skin and soft tissue toxicity : Grade 2 | 27
  Late skin and soft tissue toxicity : Grade 1 | 34
  Late skin and soft tissue toxicity : Grade 2 | 3

ADVERSE EVENTS:
Description: Serious Adverse Events and Other Adverse Events were not collected/assessed.
Arm/Group | Active Breathing Coordinator
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes